CLINICAL TRIAL: NCT02022735
Title: Deep Brain Stimulation Effects on Gait and Balance in Patients With Parkinson's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding not secured
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Corneliu C Luca, Assistant Professor of Neurology, University of Miami
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 20130225
Record Dates: First submitted 2013-12-05; First posted 2013-12-30 (Estimated); Results first posted 2021-04-01 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Parkinson's Disease
Keywords: Deep Brain Stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Bilateral stimulation (Experimental): Participants will receive Deep Brain Stimulation Bilaterally.
  Interventions: Device: Deep Brain Stimulator
- Left stimulation (Experimental): Participants will receive Deep Brain Stimulation on the left side only
  Interventions: Device: Deep Brain Stimulator
- Right stimulation (Experimental): Participants will receive Deep Brain Stimulation on the right side only
  Interventions: Device: Deep Brain Stimulator
- Off stimulation (No Intervention): Participants will receive no brain stimulation

INTERVENTIONS:
Device: Deep Brain Stimulator — DBS will provide brain stimulation.
  Other Names: DBS
  Arms: Bilateral stimulation; Left stimulation; Right stimulation

SUMMARY:
The purpose of this study is to evaluate the effect of Deep Brain stimulation (DBS) on walking in patients with Parkinson's disease that have had DBS. While DBS improves Parkinson's disease (PD) symptoms and walking in many patients in some of the patients walking problems persist. This study aims to find out what are the best stimulation parameters of the DBS in order to improve walking.

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic Parkinson's disease stage 1-3 that underwent subthalamic nucleus (STN) Deep Brain Stimulation (DBS) and have walking difficulties 6-12 months after DBS.
* On stable dose of dopaminergic drugs
* Age 45-70 years of age

Exclusion Criteria:

* Past medical history of seizures
* Renal insufficiency
* Cardiac arrhythmia
* Severe arthritis
* Women of childbearing potential
* Dementia
* Less than 45 years of age or older than 70 years of age

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-09-01; Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corneliu Luca, MD, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: All participants enrolled in the study completed the 4 arms crossover study design. All participants received and was evaluated for all four interventions: Bilateral Deep Brain Stimulation (DBS), Right Side DBS, Left side DBS and Off/No Stimulation.
Period: Overall Study
Arm/Group | All Participants
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants that completed the 4 arm crossover study design
Arm/Group | All Participants
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 13

OUTCOME MEASURES:

1. Primary Outcome: Walking Speed
Description: Walking speed will be measured using sensors reported in meter per second.
Time Frame: Up to 1 hour
Population: All participants completed all 4 arms in the cross over study design.
Measure: Mean (Standard Deviation); unit: meter per second
Groups:
- OFF Stimulation: Participants will receive no Deep Brain Stimulation
Arm/Group | Bilateral Stimulation | Left Stimulation | Right Stimulation | OFF Stimulation
Number analyzed (Participants) | 22 | 22 | 22 | 22
meter per second | 0.95 (0.05) | 0.90 (0.05) | 0.92 (0.05) | 0.84 (0.07)

2. Secondary Outcome: Stride Length
Description: Stride length will be measured using sensors and will be reported in meters.
Time Frame: Up to 1 hour
Population: all participants completed all 4 arms in the crossover study design.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Bilateral Stimulation | Left Stimulation | Right Stimulation | OFF Stimulation
Number analyzed (Participants) | 22 | 22 | 22 | 22
meters | 1.09 (0.04) | 1.01 (0.05) | 1.06 (0.04) | 0.95 (0.06)

3. Secondary Outcome: UPDRS Scores
Description: Unified Parkinson's disease rating Scale (UPDRS) has a total score ranging from 0-108 with the highest score indicating worse condition.
Time Frame: Up to 1 hour
Population: All participants completed all 4 arms in the crossover study design
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bilateral Stimulation | Left Stimulation | Right Stimulation | OFF Stimulation
Number analyzed (Participants) | 22 | 22 | 22 | 22
score on a scale | 24.09 (2.76) | 38.36 (3.52) | 35.59 (3.19) | 48.68 (3.41)

4. Secondary Outcome: TUG Test
Description: Time Up and Go (TUG) Test reports the time it takes for participant to stand up from chair, walk around a cone and return to chair.
Time Frame: Up to 1 hour
Population: Team member with access to TUG score data analysis has left the institution. PI was not given access to retrieve data prior to study team member leaving the institution.
Arm/Group | Bilateral Stimulation | Left Stimulation | Right Stimulation | OFF Stimulation
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 7 hours
Arm/Group | Bilateral Stimulation | Left Stimulation | Right Stimulation | OFF Stimulation
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22 | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-04): https://cdn.clinicaltrials.gov/large-docs/35/NCT02022735/Prot_SAP_000.pdf